CLINICAL TRIAL: NCT02403817
Title: Wireless EEG System for Training Attention and Eye Movement in ASD
Brief Title: Training Attention and Eye Movement in ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jeanne Townsend, PhD, Professor of Neurosciences, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R33MH096967 (NIH)
Record Dates: First submitted 2015-03-23; First posted 2015-03-31 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Autistic Disorder; Autism Spectrum Disorder
Keywords: Video Games
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: This project develops the intervention and includes a small clinical (behavioral) trial for ASD participants. A small number of ASD participants will be randomly assigned to intervention 'games' played by mouse response--the others to gaze-driven response.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye Movement Game Control (Experimental): Cognitive Training Eye Motor Training
  Interventions: Behavioral: Cognitive Training; Behavioral: Eye Motor Training
- Hand Movement Game Control (Active Comparator): Cognitive Training Hand Motor Training
  Interventions: Behavioral: Cognitive Training; Behavioral: Hand Motor Training

INTERVENTIONS:
Behavioral: Cognitive Training — A collection of video games that rely on various aspects of visual behavior (i.e. sustained attention, vigilance, rapid discrimination, etc) for successful play.
Behavioral: Eye Motor Training — Game play will be controlled by the player's eye movements (via an eye tracking device)
  Arms: Eye Movement Game Control
Behavioral: Hand Motor Training — Game play will be controlled by the player's hand movements (via a joystick).
  Arms: Hand Movement Game Control

SUMMARY:
Current therapies for autism target social and language behaviors, but due to the high-level nature of these skills any improvement rarely extends beyond the targeted behavior. This project uses new technology to implement a novel concept for behavioral intervention to improve basic attention and eye movement skills in ASD. Because these basic skills form the foundation for good social communication, training these abilities has the potential to improve a broad spectrum of clinical symptoms, and in young children may affect the course of development.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a lifelong disorder that severely affects the ability to learn and function in a social environment. In typical function, higher level social, language and communication skills develop over the first few years of life and depend upon the critical building blocks of sensory-motor and attention abilities. Similarly in autism, higher level problems with social communication develop over the first two post-natal years and are preceded by subtle but abnormal visual attention and motor skills. Trainings to improve social interaction and communication are the most common of behavioral interventions in ASD. These therapies may improve the specific behaviors that are targets of the training, but rarely do they generalize to broader function or other clinical symptoms. The investigators propose that interventions aimed instead at the early deficits that support social and language skills would be more broadly effective. Because disruption of attention is one of the earliest and most persistent symptoms in autism, and because attention is highly subject to improvement with training, it is an important target for intervention.

This a novel intervention to train the speed and accuracy of attention orienting and eye movement. The training is designed to target attentional behaviors that have been shown to be impaired in autism, including attention orienting, disengagement and shifting, and a restricted attentional field. Because eye movement and attention are tightly linked, eye movement deficits in ASD parallel those found in spatial attention. Eye movements provide a marker for attention and the proposed training is designed to improve speed, accuracy and flexibility of eye movement and attention simultaneously. Training uses a series of entertaining video games to gradually shape behavior using visual and auditory feedback provided in real time. The investigators plan three levels of outcome measures for pre- and post-training to test the effectiveness of the intervention (direct tests of attention and eye movement; tests of improvement in attentional and visual monitoring and speed and accuracy of response in a simulated environment; tests of behavior in an actual social environment). The investigators will conduct clinical trials with control conditions (e.g., standard video games without training elements) with a small sample of ASD children aged 9-15. If this initial work is successful, the long term goal is to develop a readily available inexpensive eyetracker-based system for home use that is suitable for a broad age range of ASD children and adults.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of Autism Spectrum Disorder (on Diagnostic and Statistical Manual -IV, Autism Diagnostic Observation Schedule, Autism Diagnostic Interview-Revised)
* Participant has a nonverbal Intelligence Quotient (IQ) of 85 or greater and verbal IQ of 70 or greater
* Cooperative and able to follow instructions
* Normal hearing acuity
* Normal or corrected-to-normal vision

Exclusion Criteria:

* Major medical or neurological problems including seizures, diagnosed epileptiform EEG abnormalities, migraine, tuberous sclerosis, fragile X, static encephalopathies resulting from prior Central Nervous System insults, significant premature birth, and history of exposure to teratogens, metabolic abnormalities, and history of head trauma, cerebral palsy, stroke, meningitis, brain tumor or additional psychiatric diagnoses
* Participants currently participating in vision therapy will be excluded

Ages: 9 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Townsend, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD is being shared through National Institutes of Health (NIH) National Database for Autism Research (NDAR).
Time Frame: Data are available to share now (August 8, 2019) and can remain available indefinitely or as long as the National Database for Autism Research is supported.
Access Criteria: Data are shared through the National Database for Autism Research. Access is by registration and meeting eligibility requirements established by the National Institutes of Health for data sharing.

RESULTS

PARTICIPANT FLOW:
Groups:
- Eye Movement Game Control: Cognitive Training Eye Motor Training
  Cognitive Training: A collection of video games that rely on various aspects of visual behavior (i.e. sustained attention, vigilance, rapid discrimination, etc) for successful play.
  Eye Motor Training: Gameplay will be controlled by the player's eye movements (via an eye tracking device)
- Hand Movement Game Control: Cognitive Training Hand Motor Training
  Cognitive Training: A collection of video games that rely on various aspects of visual behavior (i.e. sustained attention, vigilance, rapid discrimination, etc) for successful play.
  Hand Motor Training: Gameplay will be controlled by the player's hand movements (via a joystick).
Period: Overall Study
Arm/Group | Eye Movement Game Control | Hand Movement Game Control
Started | 28 | 2
Completed | 23 | 2
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Population: These are the participants that completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eye Movement Game Control | Hand Movement Game Control | Total
Number analyzed (Participants) | 23 | 2 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.31 (4.3) | 21.41 (.4) | 17.62 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 18 | 2 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 2 | 14
  More than one race | 7 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 2 | 25
Autism Diagnosis [Count of Participants; unit: Participants] | 23 | 2 | 25

OUTCOME MEASURES:

1. Primary Outcome: Spatial Attention Baseline
Description: This behavioral task assesses the participant's baseline ability to rapidly and accurately shift visual attention to different spatial locations. This task also reveals whether a participant becomes overly-focused ('stuck') at specific locations.
Time Frame: Pre-intervention
Population: All participants who completed the 8 weeks of game-based training were analyzed.
Measure: Mean (Standard Deviation); unit: Percent Correct
Arm/Group | Eye Movement Game Control | Hand Movement Game Control
Number analyzed (Participants) | 23 | 2
Percent Correct | 80.3 (14.8) | 43.0 (26.9)

2. Primary Outcome: Saccadic Eye Movements Baseline
Description: This task uses an eyetracker to measure the baseline speed and accuracy of a participant's saccadic eye movements in response to various stimuli. Measure is accuracy of first saccade in the anti-saccade task.
Time Frame: Pre-intervention
Population: Because of technical difficulties we have only partial data for this measure.
Measure: Mean (Standard Deviation); unit: percent correct direction
Arm/Group | Eye Movement Game Control | Hand Movement Game Control
Number analyzed (Participants) | 16 | 0
percent correct direction | 49.20 (2.8) |

3. Primary Outcome: Change in Spatial Attention at 8 Weeks
Description: This behavioral task assesses the change in the participant's ability to rapidly and accurately shift visual attention to different spatial locations as a result of the intervention.
Time Frame: end of Week 8
Population: All participants who completed 8 weeks of training were analyzed.
Measure: Mean (Standard Deviation); unit: Percent Correct
Arm/Group | Eye Movement Game Control | Hand Movement Game Control
Number analyzed (Participants) | 23 | 2
Percent Correct | 88.07 (13.9) | 77.5 (16.3)
Statistical Analysis 1: Comparison: Eye Movement Game Control; This analysis compares pre-intervention to post-intervention scores in the eye movement training group on the primary attention outcome measure. The hand movement Control in this pilot was not feasible and the sample is too small for analysis. This is a small pilot study and so power analyses were not computed. The null hypothesis was no difference between pre- and post-training outcome measure (alpha .05); Test type: Other — This is a small pilot study with no power calculations required (and no data upon which to base a priori power estimates); p = 0.00005, t-test, 2 sided

4. Primary Outcome: Change in Saccadic Eye Movements at 8 Weeks
Description: This task uses an eyetracker to measure the change in the speed and accuracy of a participant's saccadic eye movements in response to various stimuli as a result of the intervention. Measure is accuracy of first saccade in an anti-saccade task.
Time Frame: end of Week 8
Population: Because of technical difficulties we have data for only part of the sample.
Measure: Mean (Standard Deviation); unit: Percent Correct Direction
Arm/Group | Eye Movement Game Control | Hand Movement Game Control
Number analyzed (Participants) | 16 | 0
Percent Correct Direction | 59.4 (2.7) |
Statistical Analysis 1: Comparison: Eye Movement Game Control; This analysis compares pre-intervention to post-intervention scores in the eye movement training group on the primary eye movement outcome measure. The hand movement Control in this pilot was not feasible and the sample is too small for analysis. This is a small pilot study and so power analyses were not computed. The null hypothesis was no difference between pre- and post-training outcome measure (alpha .05); Test type: Other; p = 0.018, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: For each subject, data were collected from initial enrollment for 8 weeks.
Description: Definition not different.
Arm/Group | Eye Movement Game Control | Hand Movement Game Control
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/2
Other Adverse Events (participants affected / at risk) | 0/28 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT02403817/Prot_SAP_000.pdf